CLINICAL TRIAL: NCT06386302
Title: A Multicenter, Randomized, Controlled Clinical Trial of Chidamide Combined With Venetoclax and Azacitidine in the Treatment of Newly Diagnosed Acute Myeloid Leukemia (AML) Who Are Not Suitable for Intensive Chemotherapy
Brief Title: Chidamide, Venetoclax, and Azacitidine for Newly Diagnosed Acute Myeloid Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023074
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-12

CONDITIONS: AML; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chidamide combined with venetoclax, azacitidine group (Experimental): Chidamide (C): 30 mg/d orally on d1, 4, 8, 11 or 10 mg QD, d1-d14, adjusted according to patient tolerance Azacitidine (A): 75 mg/m 2 /d subcutaneous injection d1-d7 Venetoclax (V): 100 mg d1 200 mg d 2 400 mg d3-d28 Orally
  A treatment cycle is 28 days , and subjects will continue to receive treatment allocation according to the investigator's assessment until documented disease progression, intolerable toxicity, withdrawal of consent, or the subject meets other conditions for terminating treatment. Program Standards (whichever occurs first).
  Interventions: Drug: Chidamide; Drug: Venetoclax; Drug: azacitidine
- venetoclax, azacitidine group (Active Comparator): azacitidine: 75 mg/m 2 /d subcutaneous injection d1-d7 Venetoclax: 100 mg day 1, 200 mg day 2, 400 mg day 3-d28 orally A treatment cycle is 28 days , and subjects will continue to receive treatment allocation according to the investigator's assessment until documented disease progression, intolerable toxicity, withdrawal of consent, or the subject meets other conditions for terminating treatment. Program Standards (whichever occurs first).
  Interventions: Drug: Venetoclax; Drug: azacitidine

INTERVENTIONS:
Drug: Chidamide — 30 mg/d orally twice-weekly
  Arms: Chidamide combined with venetoclax, azacitidine group
Drug: Venetoclax — 100 mg d1 200 mg d 2 400 mg d3-d28 Orally
Drug: azacitidine — 75 mg/m 2 /d subcutaneous injection or IV d1-d7

SUMMARY:
To evaluate the feasibility, effectiveness and safety of chidamide combined with venetoclax and azacitidine in the treatment of newly diagnosed acute myeloid leukemia (AML) who are not suitable for intensive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* （1）Age ≥18 years old, no gender limit ;
* （2）be diagnosed with AML (non-M3) according to WHO 2016 standards;
* （3）No previous treatment;
* （4）Ineligible for intensive chemotherapy based on the following definitions: ≥75 years of age or 18 to 74 years of age with at least one of the following comorbidities: Eastern Cooperative Oncology Group (ECOG) performance status of 2 or 3 A history of cardiac disease such as congestive heart failure Treatment is required, or ejection fraction ≤ 50%, or chronic stable angina, diffusing capacity of lung for carbon monoxide (DLCO) ≤ 65%, or forced expiratory volume in first second (FEV1) ≤ 65%, creatinine clearance ≥ 30 mL/min to < 45 mL/min, moderate hepatic impairment, total bilirubin > 1.5 to ≤ 3.0 × ULN, other comorbidities that are not suitable for intensive chemotherapy in the physician's judgment.
* （5）Subjects must have an ECOG performance status score of: 0 to 2 for subjects aged ≥ 75 years or 0 to 3 for subjects aged ≥ 18 to 74 years.
* （6）Other comorbidities that are not suitable for intensive chemotherapy in the doctor's judgment;
* （7）Expected survival time ≥3 months;
* （8）Have the ability to understand and be willing to sign the informed consent form for this study.

Exclusion Criteria:

* (1) Combined with other malignant tumors
* (2) Have ever received treatment with chidamide and / or venetoclax or azacitidine;
* (3) The risk is assessed as low risk according to the NCCN 2022 guidelines [t(8;21)(q22;q22.1);RUNX1-RUNX1T1, inv(16)(p13.1q22) or t(16;16 )(p13.1;q22);CBFB-MYH11 ] ;
* (4) The subject is known to have AML central nervous system (CNS) infiltration;
* (5) Have undergone cardiac angioplasty or stent placement within 12 months before signing the informed consent form , or have a history of myocardial infarction, unstable angina, or other clinically significant heart disease;
* (6 ) Active infections (including bacterial, fungal or viral infections) and organ bleeding that cannot be controlled clinically;
* (7) Pregnant or lactating women;
* (8) Participated in any other clinical research within 3 months before signing the informed consent form ;
* (9 ) The researcher believes that it is not suitable to participate in this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission rate | 2 months
  Composite complete remission rate after 2 cycles of treatment [Complete remission, CR) + complete remission with incomplete blood count (CR with incomplete blood count recovery, CRi); CR + CRi ]

SECONDARY OUTCOMES:
Overall response rate (ORR) | 24months
  Overall response rate (ORR), including complete remission (Complete remission (CR), complete remission with incomplete blood count (CR with incomplete blood count recovery (CRi), morphological leukemia free state (MLFS), and partial remission (PR) as a percentage of the total number of patients participating in the efficacy analysis.
Overall survival (OS) | 24months
  Overall survival (OS): defined as the number of days from the date of randomization to the date of death. Subjects who have not died will be censored on the last date they are known to be alive .
MRD response rate | 24months
  Minimal residual disease (MRD)rate: defined as less than 0.1% remaining blasts per white blood cell, as measured by bone marrow examination. Other thresholds can also be explored and correlated with efficacy results. Subjects who are randomized but not assessed for MRD will be considered MRD response rate non-responders. The proportion of subjects achieving an MRD response (CR + CRi) was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, MD, Principal Investigator — Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Blood Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No